CLINICAL TRIAL: NCT02869373
Title: Assistant Professor
Brief Title: Spinal Stabilization Exercise Effects in Hypermobility
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, Assistant Professor, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015-64/82
Record Dates: First submitted 2016-08-12; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Hypermobility Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor

ARMS (2):
- Exercise (Experimental): spinal stabilization exercise program was applied
  Interventions: Behavioral: spinal stabilizaton exercise
- Control (No Intervention)

INTERVENTIONS:
Behavioral: spinal stabilizaton exercise — In Exercise group, spinal stabilization exercise program was carried out 3 days a week for 8 weeks.
  Arms: Exercise

SUMMARY:
The aim of this study is to investigate the effects of an 8-week lumbar spinal stabilization exercise program on pain, trunk muscle endurance and postural stability in women with benign joint hypermobility syndrome

ELIGIBILITY:
Inclusion Criteria:

* volunteers in an age range of 18 to 30,
* being women,
* having benign joint hypermobility syndrome diagnosed according to the Brighton criteria,
* having no contraindication to join an exercise program.

Exclusion Criteria:

* having rheumatologic or neurologic diseases,
* any other pathology involving the musculoskeletal system-history of fractures, joint dislocations, sprains and strains,
* associated connective tissue disorders including Marfan syndrome, Ehlers-Danlos syndrome, osteogenesis imperfecta,
* severe psychological disorders,
* being pregnant,
* intervention including exercise or physical therapy in the last 3 months.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in musculoskeletal pain intensity as measured by Visual Analog Scale | Change from baseline musculoskeletal pain intensity at 8 weeks

SECONDARY OUTCOMES:
Change in trunk muscle endurance as measued with McGill's trunk muscle endurance tests | Change from baseline trunk muscle endurance at 8 weeks
Change in postural stability as measured with Biodex Balance System SD | Change from baseline postural stability at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Seyda TOPRAK CELENAY, Study Director — Ankara Yildirim Beyazıt University; Derya OZER KAYA, Principal Investigator — Izmir Katip Celebi University